CLINICAL TRIAL: NCT04137601
Title: Congenital Syphilis at Third-level Pediatric Hospital. A Prospective Cohort With Retrospective Evaluation Study of the Last Three Decades.
Brief Title: Congenital Syphilis Prospective Cohort With Retrospective Evaluation
Status: Completed | Type: Observational
Sponsor: Hospital de Niños R. Gutierrez de Buenos Aires (Other)
Responsible Party: Principal Investigator, Dr Jaime Altcheh, Principal Investigator, Hospital de Niños R. Gutierrez de Buenos Aires
Other Study IDs: SiC cohort
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Syphilis, Congenital
Keywords: Congenital syphilis; VDRL; CSF; Clinical manifestations
MeSH Terms: conditions — Syphilis, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Syphilis is an infectious disease caused by Treponema pallidum. In children, there are two different forms of this disease; acquired syphilis and congenital syphilis, which results from transplacental transmission of spirochetes.

The worldwide incidence of congenital syphilis has increased in past years, probably due to inadequate control of pregnant women and lack of early diagnose and treatment in acute infected adults.

This infection can have numerous and non-specific manifestations at all stages, and may simulate other diseases, which can delay diagnose if not suspected.

A high number of newborns can be asymptomatic, so diagnose is confirmed or discharged by serologic testing after 6 to 10 months of age.

This study will observe the clinical presentation and the laboratory of patients with CS treated.

ELIGIBILITY:
Inclusion Criteria:

* Infants with reactive VDRL /RPR of mothers with positive serology without confirmed treatment or incomplete.
* Patients with compatible clinical signs of syphils.

Exclusion Criteria:

* Patients with diagnosis of acquired syphilis
* Patients whose medical records are missing

Ages: 0 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In older children, the sexual route for abuse will be ruled out as a means of interrogation infection and analysis of family dynamics by a multidisciplinary team.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Analyze the number of cases of congenital syphilis according to the years surveyed at the Ricardo Gutierrez Children's Hospital | Past 30 years
  By examining clinical records we will describe prevalence of congenital syphilis through last 30 years.

SECONDARY OUTCOMES:
Describe the clinical presentation -symptoms and image findings - in children diagnosed with CS. Symptoms will be measured as present or not and described. | Past 30 years
  By looking at clinical records we will describe the number of children presenting with symptoms and number of asymptomatic. We will also describe the most frequent symptoms found and other test findings.

OTHER OUTCOMES:
Estimate the most frequent laboratory alterations in patients with CS | Past 30 years
  By analizing clinical records we will describe the laboratory findings in both symptomatic and asymptomatic children with CS.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Altcheh, Dr, Principal Investigator — Principal Investigator
Locations (1):
- Parasitology Division, Children's Hospital "R Gutierrez" of Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided